CLINICAL TRIAL: NCT00982319
Title: Evaluating the Effect of Broccoli Sprouts (Sulforaphane) on Cellular Proliferation, an Intermediate Marker of Breast Cancer Risk
Brief Title: Study to Evaluate the Effect of Sulforaphane in Broccoli Sprout Extract on Breast Tissue
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: J0822
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Results first posted 2018-07-31 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Breast Cancer
Keywords: Broccoli Sprout Extract; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Broccoli sprout extract (Experimental): Patients will be randomized to 14 day intervention of broccoli sprout extract and mango juice consisting of a dose of 100 µmols of sulforaphane dissolved in 150 mL mango juice once a day.
  Interventions: Drug: Broccoli sprout extract; Drug: Mango juice
- Mango juice (Placebo Comparator): Patients will be randomized to 14 day intervention of 150 mL mango juice without broccoli sprout extract extract once a day.
  Interventions: Drug: Mango juice

INTERVENTIONS:
Drug: Broccoli sprout extract — 100 µmols of sulforaphane (dissolvable)
  Arms: Broccoli sprout extract
Drug: Mango juice — 150 mL of mango juice

SUMMARY:
The purpose of this research is to examine the effect of a broccoli sprout preparation on specific factors in breast tissue that are related to breast cancer risk and to assess whether sulforaphane a key component of broccoli sprouts increases the levels of protective enzymes in breast tissue. In addition, the investigators will also examine how acceptable the broccoli sprouts preparation is to the study participants.

DETAILED DESCRIPTION:
A double-blind randomized Phase II chemoprevention trial of BSE versus placebo will be conducted in up to 35 women diagnosed with DCIS on core biopsy prior to their definitive surgery (study diagram below). The primary study endpoint will be a decrease in the mean proliferative rate measured by Ki67%.

Women diagnosed with DCIS on core or incisional/excisional biopsy scheduled for definitive surgery at Johns Hopkins Hospital will be recruited for this study. Participants will be placed on a cruciferous free diet for the 14 days prior to their surgical date and drink a randomized intervention beverage (mango juice with or without broccoli sprout extract). Additionally participants will provide 2 blood and 2 urine sample collections, report medication use and adverse events using prepared forms and complete a daily diet check list during the 14 day intervention. On the day of definitive breast surgery, 1-2 grams of breast tissue (including normal adjacent breast tissue) will be collected during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female 18 + years of age
* Confirmed diagnosis of DCIS on core or excisional/incisional biopsy and scheduled for definitive surgery
* Pre or Post menopausal women reporting no use of hormone replacement therapy, tamoxifen or raloxifene within the prior 6 months to eligibility screening
* Agree to avoid cruciferous vegetable/condiment intake for 14 days
* Agree to sign an informed consent and allow use of some tissue (slides) from biopsy and definitive surgery for research purposes

Exclusion Criteria:

* Prior cancer diagnosis other than non-melanomatous skin cancer or cervical carcinoma in-situ
* Used hormone replacement therapy, tamoxifen or raloxifene within the past 6 months prior to eligibility screening
* Used antibiotics within 10 days prior to beginning cruciferous free diet (day -14 prior to surgery)
* Smoked within the past 12 months prior to eligibility screening;
* Active infection or inflammation of the breast at time of eligibility screening
* Has baseline comprehensive metabolic panel (CMP) [Glucose, Calcium, Albumin, Serum total protein (TP), Sodium, Potassium, Carbon dioxide, Chloride, Blood urea nitrogen (BUN), Creatinine, Alkaline phosphatase (ALP), Alanine amino transferase (AST), Aspartate amino transferase (SGOT), and Bilirubin], prothrombin time (PT) and , complete blood count (CBC) values that are 1.5 times in either direction the reported normal range

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kala Visvanathan, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health and Sidney Kimmel Comprehensive Cancer Center
Locations (1):
- Johns Hopkins Medical Institution, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Broccoli Sprout Extract and Mango Juice: Patients will be randomized to 14 day intervention of broccoli sprout extract consisting of a consistent dose of sulforaphane dissolved in mango juice compared to a placebo preparation of mango juice alone. All women will be on a cruciferous free diet for the duration of the study (14 days).
  Broccoli sprout extract (sulforaphane): Women newly diagnosed with DCIS on core biopsy prior to definitive surgery will be randomized to receive a prepartion of broccoli sprout extract and mango juice. All women will be on a cruciferous free diet for the duration of the study (14 days) and complete a daily dietary check list. Twelve hour urine collections and blood samples will be collected at various time points during the study. Acceptability of the 14 day dose will be evaluated by monitoring indices of compliance, including urinary measurements of ITC excretion, the daily food check list and a questionnaire administered at the end of the study.
- Mango Juice: Patients will be randomized to 14 day intervention of mango juice without broccoli sprout extract. All women will be on a cruciferous free diet for the duration of the study (14 days).Mango juice without extract: Mango juice without broccoli sprout extract.
  B Mango juice: Women newly diagnosed with DCIS on core biopsy prior to definitive surgery will be randomized to receive a placebo preparation of mango juice alone. All women will be on a cruciferous free diet for the duration of the study (14 days) and complete a daily dietary check list. Twelve hour urine collections and blood samples will be collected at various time points during the study. Acceptability of the 14 day dose will be evaluated by monitoring indices of compliance, including urinary measurements of ITC excretion, the daily food check list and a questionnaire administered at the end of the study.
Period: Overall Study
Arm/Group | Broccoli Sprout Extract and Mango Juice | Mango Juice
Started | 17 | 17
Completed | 15 | 15
Not Completed | 2 | 2
Not completed — Surgery date change | 1 | 0
Not completed — Preop values out of acceptable range | 1 | 1
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Broccoli Sprout Extract and Mango Juice: Patients will be randomized to 14 day intervention of broccoli sprout extract consisting of a consistent dose of sulforaphane dissolved in mango juice compared to a placebo preparation of mango juice alone. All women will be on a cruciferous free diet for the duration of the study (14 days).
  Broccoli sprout extract (sulforaphane): Women newly diagnosed with DCIS on core biopsy prior to definitive surgery will be randomized to either a prepartion of broccoli sprout extract and mango juice or a placebo preparation of mango juice alone. All women will be on a cruciferous free diet for the duration of the study (14 days) and complete a daily dietary check list. Twelve hour urine collections and blood samples will be collected at various time points during the study. Acceptability of the 14 day dose will be evaluated by monitoring indices of compliance, including urinary measurements of ITC excretion, the daily food check list and a questionnaire administered at the end of the study.
- Mango Juice: Patients will be randomized to 14 day intervention of Mango juice without broccoli extract. All women will be on a cruciferous free diet for the duration of the study (14 days).
  Mango juice: Women newly diagnosed with DCIS on core biopsy prior to definitive surgery will be randomized to either a prepartion of broccoli sprout extract and mango juice or a placebo preparation of mango juice alone. All women will be on a cruciferous free diet for the duration of the study (14 days) and complete a daily dietary check list. Twelve hour urine collections and blood samples will be collected at various time points during the study. Acceptability of the 14 day dose will be evaluated by monitoring indices of compliance, including urinary measurements of ITC excretion, the daily food check list and a questionnaire administered at the end of the study.
- Total: Total of all reporting groups
Arm/Group | Broccoli Sprout Extract and Mango Juice | Mango Juice | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants] — Age collected on baseline survey. Participants had to be 18+ years old
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 13 | 12 | 25
    >=65 years | 2 | 3 | 5
Age, Continuous [Median (Full Range); unit: years] | 52 [35 to 71] | 54 [40 to 72] | 53 [35 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Mean Proliferative Rate Measured by Ki67%
Description: Pathologists score the slides without knowledge of treatment assignment at the end of the study. All pre-post samples from one individual will be evaluated together. Quality control for these stains is performed routinely in the immunohistochemistry lab (using lymphoid tissue for Ki67). Initial scoring is performed where possible on a minimum of 3000 cells, by counting the number of positive cells divided by the total number of cells. DCIS lesions will be scored separately to adjacent normal tissue. The rationale for selecting Ki67 as a measure of cellular proliferation includes the robustness of the staining reaction, correlation with the S phase fraction of the cell cycle and mitotic index and that it can be successfully ascertained from core breast biopsies provided there is an adequate yield of epithelial cells. A negative value reflects a decrease in ki67 positive cells, therefore a decrease in cellular proliferation.
Time Frame: Change from baseline to 14 days post-intervention
Population: All participants who completed the 14-day intervention on either study arm were included in analysis.
Measure: Mean (Standard Deviation); unit: percentage of Ki67
Groups:
- Broccoli Sprout Extract and Mango Juice: Patients will be randomized to 14 day intervention of broccoli sprout extract consisting of a consistent dose of sulforaphane dissolved in mango juice. All women will be on a cruciferous free diet for the duration of the study (14 days).
- Mango Juice Without Extract: Patients will be randomized to 14 day intervention of mango juice alone. All women will be on a cruciferous free diet for the duration of the study (14 days).
Arm/Group | Broccoli Sprout Extract and Mango Juice | Mango Juice Without Extract
Number analyzed (Participants) | 15 | 15
percentage of Ki67 | -1.15 (2.08) | 4 (17.08)
Statistical Analysis 1: Comparison: Broccoli Sprout Extract and Mango Juice vs Mango Juice Without Extract; Test type: Superiority; p = 0.32, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Phase II Protein Expression as Assessed by Change in Cytoprotective Enzyme Expression Within Tumor
Description: Phase II protein expression of cytoprotective enzymes known to be modulated by sulforaphane in DCIS specimens.
  Cytoprotective enzymes measured (NQ01 and AKR1C1 expression) based on immunohistochemical analysis. Expression was categorized by the study pathologist based on percentage of cells expressing antibody on the slide.
Time Frame: Change from baseline to 14 days post-intervention
Measure: Mean (Standard Deviation); unit: % change of expression in tumor cells
Arm/Group | Broccoli Sprout Extract and Mango Juice | Mango Juice Without Extract
Number analyzed (Participants) | 15 | 15
% change of expression in tumor cells
  AKR1C1 | 62.1 (312.99) | 867.4 (2097.8)
  NQO1 | 730.98 (2411.96) | 6.34 (30.12)

ADVERSE EVENTS:
Time Frame: 14 days during the intervention period (prior to first and 3 times during intervention)
Arm/Group | Broccoli Sprout Extract and Mango Juice | Mango Juice
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 9/15 | 9/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Broccoli Sprout Extract and Mango Juice (N=15) | Mango Juice (N=15)
constipation (Gastrointestinal disorders) | 5 (9) | 4 (7)
intestional gas/bloating (Gastrointestinal disorders) | 4 (6) | 2 (6)
upset stomach/indigestion (Gastrointestinal disorders) | 1 (1) | 1 (1)
nausea/vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0)
abdominal cramps (Gastrointestinal disorders) | 0 (0) | 2 (2)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
appetite/ taste alteration (Gastrointestinal disorders) | 2 (2) | 1 (1)
light headed/ mild anxiety (Nervous system disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Eligible patients had to have their definitive breast cancer surgery at Johns Hopkins Hospital

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No